CLINICAL TRIAL: NCT05135052
Title: Efficacy of Personalised Irradiation With Rhenium-Skin Cancer Therapy (SCT) for the Treatment of Non-Melanoma Skin Cancer: A Phase IV, Multi-Centre, International, Open-Label, Single Arm Study.
Brief Title: Rhenium-Skin Cancer Therapy (SCT) for the Treatment of Non-Melanoma Skin Cancer.
Acronym: EPIC-Skin
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OncoBeta Therapeutics (Industry)
Responsible Party: Sponsor
Organization: OncoBeta International GmbH (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OB-RHSCT-101
Record Dates: First submitted 2021-10-08; First posted 2021-11-26 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Non-melanoma Skin Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Treatment with Rhenium-SCT, Single treatment.
  Interventions: Device: Rhenium-SCT

INTERVENTIONS:
Device: Rhenium-SCT — Rhenium-SCT irradiation device

SUMMARY:
Efficacy of Personalised Irradiation with Rhenium-Skin Cancer Therapy (SCT) for the treatment of non-melanoma skin cancer; a phase IV multi-centre, international, open label, single arm study.

ELIGIBILITY:
Inclusion Criteria:

1. Stage I or II BCC or SCC (SCC Well to Moderately Differentiated), and clinically node negative disease
2. Confirmed Histology, and with depth of lesion noted
3. Subjects with up to 3 lesions suitable to enter the study (subjects with more than 3 lesions are not excluded from the study, however 3 target lesions are determined for study evaluation only.)
4. Subjects able and willing to comply with the requirements of the study
5. Age >=18 years
6. Informed Consent signed by the subject consenting to undergo the study
7. Lesions up to 8cm2
8. Lesions with a depth up to 3mm confirmed on biopsy report AND deemed appropriate clinically by treating clinician
9. Subjects who are not deemed suitable for surgery, for example due to tumour location, performance status or other comorbidities as deemed relevant by the treating clinician
10. Patients who may have declined Surgery and/or fractionated Radiation Therapy

Exclusion Criteria:

1. Inability to personally provide written informed consent or to understand and collaborate throughout the study
2. Inability or unwillingness to comply with study requirements
3. Prior treatment with surgery or radiation therapy for their target lesion(s)
4. Depth of lesion greater than 3mm as defined by Biopsy and/or clinical assessment
5. Lupus and Scleroderma
6. Basal cell naevus syndrome, xeroderma, vitiligo and albinism
7. Prior laser at the tumour site
8. Malignant melanoma systemic therapy ongoing
9. Any ongoing treatment for malignancy, or in the last 4 weeks prior to study entry
10. A tumour affecting nerves or bony structures
11. Clinical concern of metastatic disease
12. Pregnancy and/or Lactation
13. Pathological exclusions: Perineural Invasion, Lymphovascular invasion
14. Anatomical exclusions: NMSC's of the Medial canthus, eyelid margin (upper and lower), Vermillion lip

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2022-01-17 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) with Modified Visual RECIST tool | 12 months
  To assess the proportion of lesions achieving complete response (CR) as per MODIFIED VISUAL RECIST criteria

SECONDARY OUTCOMES:
SKINDEX-16 QoL Questionnaire | 6 months and 12 months
  The QoL questionnaire will be scored according to the author's instructions. Change from baseline in score will be calculated. Descriptive statistics will be presented for actual score and change from baseline by timepoint, overall and by tumour type (BCC/SCC).
Comfort of Treatment short questionnaire | 14 days
  Comfort of treatment assessed using a short questionnaire completed by subjects post treatment with Rhenium-SCT. The frequency (and percentage) of subjects reporting each option for each question will be presented.
cosmetic outcomes by Visual Analogue Scale | 12 months and 24 months
  Cosmetic outcome assessed by subject and Clinician, using Visual Analogue Scale. Descriptive statistics will be presented overall and by tumour type (BCC or SCC). A mixed model will be fitted with Visual Analogue Scale as the outcome variable. Tumour type and tumour stage will be included as factors. Other relevant prognostic factors assessed at Baseline will be included. From the model the adjusted mean score will be obtained and presented with 95% confidence limits. Adjusted mean score will be estimated overall and by tumour type.

OTHER OUTCOMES:
Safety as assessed by CTCAE v4.0 | 24 months
  Adverse events by severity and by relationship to Rhenium-SCT, including radiation dermatitis, dry skin, skin ulceration, alopecia, skin induration, hypo/hyperpigmentation, and telangiectasia. Adverse events will be coded using MedDRA and comprehensively summarised by System Organ Class (SOC) and Preferred Term (PT) overall, by severity and by relationship to Rhenium-SCT.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Dr Dahlhoff, MD, Study Director — Oncobeta GmbH
Locations (7):
- Australia (3):
  - Genesis Care Health Hub at RNS, Sydney, New South Wales
  - John Flynn Hospital, Tugun, Queensland
  - Hollywood Private, Perth, Western Australia
- Klinik Ottakring, Ottakring, Austria
- Rostock University Hospital, Rostock, Germany
- Steve Beko Hospital, Pretoria, South Africa
- Kings College Hospital London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided